CLINICAL TRIAL: NCT04345185
Title: Effects of Infant Egg Consumption on Child Health and Cognition Development
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Xiaozhong Wen, Principal Investigator, State University of New York at Buffalo
Other Study IDs: STUDY00004022
Record Dates: First submitted 2020-04-04; First posted 2020-04-14 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Growth & Development; Obesity; Cardiovascular Risk Factor; Metabolic Syndrome; Food Allergy; Cognitive Developmental Delay
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Project Viva: Project Viva (1999-present) enrolled 2,341 pregnancies and followed 2,128 children at delivery, 6 months, then yearly from 1 year to 15 years of child age.
  Interventions: Other: Infant egg consumption (i.e., age of introduction and frequency of intake)
- Infant Feeding Practices Study II: The Infant Feeding Practices Study II (IFPS II, 2005-2007) enrolled 3,033 pregnancies with surveys in late pregnancy, neonatal (1 month), then monthly from 2 months (N=2,552) to 12 months of infant age, and at 6 years.
  Interventions: Other: Infant egg consumption (i.e., age of introduction and frequency of intake)

INTERVENTIONS:
Other: Infant egg consumption (i.e., age of introduction and frequency of intake)

SUMMARY:
The objective of this study is to examine how infant egg consumption (age of introduction and frequency of intake) influences physical growth, obesity, cardio-metabolic health, risk of food allergy, and cognition development in mid-childhood and adolescence.

DETAILED DESCRIPTION:
The investigators will use existing data from two US longitudinal birth cohorts that tracked mother-child dyads from pregnancy to adolescence: 1) Project Viva (1999-present) that enrolled 2,341 pregnancies and followed 2,128 children at delivery, 6 months, then yearly from 1 year to 15 years of child age, and 2) the Infant Feeding Practices Study II (IFPS II, 2005-2007) that enrolled 3,033 pregnancies with surveys in late pregnancy, neonatal (1 month), then monthly from 2 months (N=2,552) to 12 months of infant age, and at 6 years. For Aim 1, the investigators will classify infants based on their age of egg introduction: never, <2 months, 2-3 months, 4-5 months, 6-8 months, 9-11 months, and 12 months. The investigators will compare physical growth, obesity, cardio-metabolic health, food allergy, and cognition test scores in mid-childhood and adolescence. The investigators will fit multi-variable linear or logistic regression models with fractional polynomial functions of the infant age of egg introduction. Both linear (e.g., earlier introduction, a higher probability of the outcome) and non-linear (e.g., threshold effect) associations will be tested. For Aim 2, The investigators will classify infants based on their frequency of egg intake: never, <once/week, once/week, 2-4 times/week, nearly daily or daily, and 2 times/day. The investigators will use similar analytic methods mentioned above to compare their later outcomes. Finally, the investigators will create an average probability of multiple child outcomes to balance across different aspects of child health and development. The investigators will identify the lowest-risk infant egg consumption when the corresponding average predicted probability of the related adverse outcomes is the lowest.

ELIGIBILITY:
Inclusion Criteria:

* Children with complete data on infant egg consumption and the corresponding health and cognition outcomes.

Exclusion Criteria:

* None.

Ages: 0 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The investigators will use existing data from two US longitudinal birth cohorts that tracked mother-child dyads from pregnancy to adolescence: 1) Project Viva (1999-present) that enrolled 2,341 pregnancies and followed 2,128 children at delivery, 6 months, then yearly from 1 year to 15 years of child age, and 2) the Infant Feeding Practices Study II (IFPS II, 2005-2007) that enrolled 3,033 pregnancies with surveys in late pregnancy, neonatal (1 month), then monthly from 2 months (N=2,552) to 12 months of infant age, and at 6 years.
Sampling Method: Non-Probability Sample
Enrollment: 5374 (Actual)
Dates: Start 1999-01-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Weight | At 6 months (infancy)
  Research staff measured children's weight in Project Viva.
Weight | 3 years (early childhood)
  Research staff measured children's weight in Project Viva.
Weight | 7 years (mid-childhood)
  Research staff measured children's weight in Project Viva.
Weight | 12-13 years (early teen)
  Research staff measured children's weight in Project Viva.
Weight | 14-15 years (mid-teen)
  Research staff measured children's weight in Project Viva.
Weight | 3 months
  In IFPS II, mothers reported infant weight in survey.
Weight | 5 months
  In IFPS II, mothers reported infant weight survey.
Weight | 7 months
  In IFPS II, mothers reported infant weight in survey.
Weight | 12 months
  In IFPS II, mothers reported infant weight in survey.
Weight | 6 years
  In IFPS II, mothers reported infant weight in survey.
Height | 6 months
  Research staff measured children's height in Project Viva.
Height | 3 years
  Research staff measured children's height in Project Viva.
Height | 7 years
  Research staff measured children's height in Project Viva.
Height | 12-13 years
  Research staff measured children's height in Project Viva.
Height | 14-15 years
  Research staff measured children's height in Project Viva.
Height | 3 months
  In IFPS II, mothers reported infant height in survey.
Height | 5 months
  In IFPS II, mothers reported infant height in survey.
Height | 7 months
  In IFPS II, mothers reported infant height in survey.
Height | 12 months
  In IFPS II, mothers reported infant height in survey.
Height | 6 years
  In IFPS II, mothers reported infant height in survey.
Waist Circumference | 6 months
  Research staff measured children's waist circumference in Project Viva.
Waist Circumference | 3 years
  Research staff measured children's waist circumference in Project Viva.
Waist Circumference | 7 years
  Research staff measured children's waist circumference in Project Viva.
Waist Circumference | 12-13 years
  Research staff measured children's waist circumference in Project Viva.
Waist Circumference | 14-15 years
  Research staff measured children's waist circumference in Project Viva.
Skinfold thickness | 3 years
  Research staff measured children's skinfold thickness in Project Viva.
Skinfold thickness | 7 years
  Research staff measured children's skinfold thickness in Project Viva.
Skinfold thickness | 12-13 years
  Research staff measured children's skinfold thickness in Project Viva.
Skinfold thickness | 14-15 years
  Research staff measured children's skinfold thickness in Project Viva.
Fat mass | 7 years
  Research staff measured children's fat mass in Project Viva.
Fat mass | 12-13 years
  Research staff measured children's fat mass in Project Viva.
Fat mass | 14-15 years
  Research staff measured children's fat mass in Project Viva.
Lean mass | 7 years
  Research staff measured children's lean mass in Project Viva.
Lean mass | 12-13 years
  Research staff measured children's lean mass in Project Viva.
Lean mass | 14-15 years
  Research staff measured children's lean mass in Project Viva.
Trunk fat mass | 7 years
  Research staff measured children's trunk fat mass in Project Viva.
Trunk fat mass | 12-13 years
  Research staff measured children's trunk fat mass in Project Viva.
Trunk fat mass | 14-15 years
  Research staff measured children's trunk fat mass in Project Viva.
Systolic blood pressure | 7 years (mid-childhood)
  Research staff measured children's systolic blood pressure in Project Viva.
Systolic blood pressure | 12-13 years (early teen)
  Research staff measured children's systolic blood pressure in Project Viva.
Systolic blood pressure | 14-15 years (mid-teen)
  Research staff measured children's systolic blood pressure in Project Viva.
Diastolic blood pressure | 7 years
  Research staff measured children's diastolic blood pressure in Project Viva.
Diastolic blood pressure | 12-13 years (early teen)
  Research staff measured children's diastolic blood pressure in Project Viva.
Diastolic blood pressure | 14-15 years (mid-teen)
  Research staff measured children's diastolic blood pressure in Project Viva.
Diagnosis of food allergy | 2 years
  Research staff measured children's food allergy in Project Viva.
Diagnosis of food allergy | 3 years
  Research staff measured children's food allergy in Project Viva.
Diagnosis of food allergy | 4 years
  Research staff measured children's food allergy in Project Viva.
Diagnosis of food allergy | 5 years
  Research staff measured children's food allergy in Project Viva.
Diagnosis of food allergy | 6 years
  Research staff measured children's food allergy in Project Viva.
Diagnosis of food allergy | 7 years
  Research staff measured children's food allergy in Project Viva.
Diagnosis of food allergy | 8 years
  Research staff measured children's food allergy in Project Viva.
Diagnosis of food allergy | 9 years
  Research staff measured children's food allergy in Project Viva.
Diagnosis of food allergy | 10 years
  Research staff measured children's food allergy in Project Viva.
Diagnosis of food allergy | 11 years
  Research staff measured children's food allergy in Project Viva.
Diagnosis of food allergy | 12-13 years (early teen)
  Research staff measured children's food allergy in Project Viva.
Diagnosis of food allergy | 14-15 years (mid-teen)
  Research staff measured children's food allergy in Project Viva.
Diagnosis of food allergy | 2 months
  In the IFPS-II mothers reported the child's food allergy.
Diagnosis of food allergy | 3 months
  In the IFPS-II mothers reported the child's food allergy.
Diagnosis of food allergy | 4 months
  In the IFPS-II mothers reported the child's food allergy.
Diagnosis of food allergy | 5 months
  In the IFPS-II mothers reported the child's food allergy.
Diagnosis of food allergy | 6 months
  In the IFPS-II mothers reported the child's food allergy.
Diagnosis of food allergy | 7 months
  In the IFPS-II mothers reported the child's food allergy.
Diagnosis of food allergy | 8 months
  In the IFPS-II mothers reported the child's food allergy.
Diagnosis of food allergy | 9 months
  In the IFPS-II mothers reported the child's food allergy.
Diagnosis of food allergy | 10 months
  In the IFPS-II mothers reported the child's food allergy.
Diagnosis of food allergy | 11 months
  In the IFPS-II mothers reported the child's food allergy.
Diagnosis of food allergy | 12 months
  In the IFPS-II mothers reported the child's food allergy.
Diagnosis of food allergy | 6 years
  In the IFPS-II mothers reported the child's food allergy.
Intelligence (PPVT-III test) | 3 years
  In Project Viva, trained research staff administered the Peabody Picture Vocabulary Test-3rd edition (PPVT-III, a test of receptive language) at 3 years of age.
Intelligence (KBIT-II test) | 7 years
  In Project Viva, trained research staff administered the Kaufman Brief Intelligence Test-2nd edition (KBIT-II, verbal and non-verbal intelligence) at 7 years of age.
Visual-motor (WRAVMA) | 3 years
  Research staff measured children's visual-motor in Project Viva. For the visual-motor domain, research staff administered the Wide Range Assessment of Visual Motor Abilities (WRAVMA) at the 3-years visit.
Visual-motor (WRAVMA) | 7 years
  Research staff measured children's visual-motor in Project Viva. At the 7-years visit, staff administered the WRAVMA visual motor (drawing) subtest only.
Memory-learning | 7 years
  Research staff measured children's memory-learning in Project Viva. For the memory-learning domain, staff administered the design memory and picture memory subsets of Wide Range Assessment of Memory and Learning (WRAML) at the 7-years visit.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Wen, Principal Investigator — State University of New York at Buffalo
Locations (1):
- Division of Behavioral Medicine Department of Pediatrics Jacobs School of Medicine and Biomedical Sciences State University of New York at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT04345185/Prot_SAP_000.pdf